CLINICAL TRIAL: NCT05694429
Title: The Effect of the Combination of Cleanser and Moisturizer Product K on Skin Rejuvenation
Brief Title: The Effect of the Combination of Cleanser and Moisturizer Product K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RMC/EC42/2022
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aesthetic; Cosmetic; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Product K cleanser and moisturizer (Experimental): Participants will used product K cleanser and moisturizer twice daily for 8 weeks
  Interventions: Other: Product K cleanser and moisturizer

INTERVENTIONS:
Other: Product K cleanser and moisturizer — Product K cleanser and moisturizer contain ingredients that may improve skin hydration and elasticity

SUMMARY:
This study is conducted to evaluate the effectiveness of product K cleanser and moisturizer when use in combination for skin rejuvenation. The study duration is 8 weeks and the skin assessment will be carried out at baseline, week 2, week 4 and week 8.The main questions this study aims to answer are:

1. The effect of cleanser and moisturizer K when use in combination on skin hydration.
2. The effect of cleanser and moisturizer K when use in combination on skin elasticity.
3. To observe any adverse effect occurrence with the usage of the products.

ELIGIBILITY:
Inclusion Criteria:

* Malaysia citizen
* Male and female (age 20-60 years old)

Exclusion Criteria:

* Participants taking isotretinoin
* Immunocompromised patients
* Participant who undergo any cosmetic procedures such as laser & light treatment for the past three months.
* Participant with a history of facial surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration from baseline and at week 2, week 4 and week 8 after using product K cleanser and moisturizer | Baseline, week 2, week 4 and week 8
  Skin hydration will be assessed using JANUS III skin analyzer
Change in skin elasticity from baseline and at week 2, week 4 and week 8 after using product K cleanser and moisturizer | Baseline, week 2, week 4 and week 8
  Skin elasticity will be assessed using JANUS III skin analyzer
Adverse effect after using product K cleanser and moisturizer | Week 8
  Based on adverse effect occurrence on participants that occur during study period (8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No